CLINICAL TRIAL: NCT00307710
Title: Evaluation of the Reactogenicity and Immunogenicity of Different Doses of Trivalent Baculovirus-expressed Influenza HA Vaccine in Adults With Non-Hodgkin's B-cell Lymphoma: A Phase II, Double-Blind Pilot Study - Version 4
Brief Title: Influenza Vaccination in Patients Receiving Antineoplastic Therapy for Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 2004-0340; DMID 04-036
Record Dates: First submitted 2006-03-24; First posted 2006-03-28 (Estimated); Last update posted 2012-07-31 (Estimated); Status verified 2012-07

CONDITIONS: Lymphoma
Keywords: Non-Hodgkin's Lymphoma; Influenza Vaccination; Trivalent Baculovirus-Expressed Influenza HA vaccine; Antineoplastic Therapy
MeSH Terms: conditions — Lymphoma; Lymphoma, Non-Hodgkin; Influenza, Human | interventions — trivalent baculovirus-expressed influenza-virus hemagglutinin vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- A: Trivalent Subvirion Vaccine (Experimental): Group A: Trivalent subvirion vaccine - standard inactivated influenza vaccine by intramuscular injection.
  Interventions: Biological: Trivalent Baculovirus-expressed Influenza HA vaccine
- B: Vaccine 15 μg (Experimental): Group B: Trivalent rHA0 vaccine 15 μg per rHA0 (total 45 μg rHA0)
  Interventions: Biological: Trivalent Baculovirus-expressed Influenza HA vaccine
- C: Vaccine 45 μg (Experimental): Group C: Trivalent rHA0 vaccine 45 μg per rHA0 (total 135 μg rHA0)
  Interventions: Biological: Trivalent Baculovirus-expressed Influenza HA vaccine
- D: Vaccine 135 μg (Experimental): Group D: Trivalent rHA0 vaccine 135 μg per rHA0 (total 405 μg rHA0)
  Interventions: Biological: Trivalent Baculovirus-expressed Influenza HA vaccine

INTERVENTIONS:
Biological: Trivalent Baculovirus-expressed Influenza HA vaccine — Receive either standard inactivated influenza vaccine or one of three doses of the experimental vaccine, vaccine dose 15, 45 or 135 μg HA per virus, intramuscular injection.

SUMMARY:
Primary Objective:

To assess the trend in immunogenic response across patients administered either licensed trivalent inactivated influenza vaccine (TIV) or one of three doses (15, 45 or 135 μg) of trivalent recombinant baculovirus expressed hemagglutinin vaccines. Immunogenic response is defined as a 4-fold or greater increase in serum antibody.

Secondary Objective:

To determine the safety and tolerability of 3 doses (15 μg HA per virus, 45 μg HA per virus, and 135 μg HA per virus) of recombinant baculovirus-expressed HA vaccine in patients with non-Hodgkin's B-cell lymphoma.

DETAILED DESCRIPTION:
Influenza is a common respiratory infection caused by viruses. Standard influenza vaccines may not be as effective at protecting cancer patients as the general population from getting influenza. New technology has been developed that allows stronger (and hopefully more effective) influenza vaccines to be developed. This research study will test an experimental influenza vaccine.

If you agree to take part in this study, you will be randomly assigned (as in the toss of a coin) to receive either standard inactivated influenza vaccine or one of three doses of the experimental vaccine. You will have an equal chance of being assigned to any of the four treatment groups. Neither your physician, the study doctor, or you will know which vaccine or dose you received. In case of an emergency, the study doctor can find out which vaccine and dose you received.

Before the injection is given, a blood test will be taken to measure your antibodies (substances that fight infection). About two teaspoons of blood will be taken for this blood test. The vaccine will be given as a one time injection in the arm. After you are given the injection, you will be observed for 20 minutes in the clinic before you are sent home. Everyone taking part in this study will be asked to keep a symptom diary and temperature log for 1 week after the injection. After 7 days, you will return for review of the diary and any symptoms you may have had.

At 4 and 8 weeks after the influenza vaccine is given, most patients will have a blood test to learn the amount of immunity against the influenza virus they have developed. About two teaspoons of blood will be required for this test. A few patients may not be eligible for the eight week blood collection and will be instructed by the study nurse about future visits to UTMDACC. Six months after you have received the vaccine, you will be contacted by one of the study personnel to ask you if you had any serious side effects that might be from the study vaccine. Once you have received this follow-up telephone call, your participation in this study will be completed.

This is an investigational study. The standard vaccine used in this study is FDA approved and commercially available. The experimental vaccine is authorized for use in research only. About 100 patients will take part in this study. All will be enrolled at UTMDACC.

This protocol is partially funded by a research contract from the National Institutes of Health (NIH) to Baylor College of Medicine.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with non-Hodgkin's B-cell lymphoma (NHL) including follicular, large cell and Mantle cell lymphoma will be included.
2. Patients in complete clinical remission and determined to have no evidence of active disease (NED).
3. Patients greater than or equal to 18 years of age who have given informed consent and signed the IRB approved informed consent.
4. Ambulatory, medically stable persons; community dwelling; able to give informed consent and available for all study visits; able to understand and comply with planned study procedures; ECOG performance status of less than or equal to 2.
5. Medically stable subjects may have underlying illnesses such as hypertension, diabetes, ischemic heart disease, or hypothyroidism, but their symptoms/signs are controlled with medical therapy.
6. Patients with a non-metastatic secondary solid tumor or malignancies not currently (< 3 months) being treated will be included.

Exclusion Criteria:

1. Patients with Hodgkin's disease, and T-cell lymphoma.
2. Patients undergoing antineoplastic therapy.
3. Patients who have received chemotherapy within the past 3 months.
4. Individuals who were given rituximab (ibritumomab tiuxetan) in < 6 months.
5. Patients receiving systemic corticosteroids and/or high-dose inhaled steroids (>800 mcg per day of beclomethasone dipropionate or equivalent).
6. Splenectomized individuals will not be included.
7. Known allergy to eggs or other components of vaccine (e.g., thimerosal).
8. Acute or chronic condition that (in the opinion of the investigator) would render vaccination unsafe or would interfere with the evaluation of responses (including but not limited to the following: acute febrile illness, known chronic liver disease; significant renal disease; oxygen-dependent chronic lung disease, New York Heart Association Functional Class III or IV dyspnea; unstable or progressive neurologic disorder; insulin-dependent diabetes mellitus).
9. Concomitant use of investigational vaccines and/or other medications within 4 weeks prior to study entry, or expected use of experimental or licensed vaccines or blood/blood products prior to study completion.
10. Previous exposure to parenteral immunoglobulins or other blood product within 6 months prior to enrollment into the study.
11. Subject is enrolled in a conflicting clinical trial.
12. Use of experimental vaccines or medications within one month of study entry.
13. Any acute or chronic condition which in the opinion of the investigator would render vaccination unsafe or interfere with the evaluation of response.
14. Patients with a known history or risk factors (IV drug abuse or casual sex within the past year) of Hepatitis B, Hepatitis C, or Human Immunodeficiency Virus.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2004-08; Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Immunogenic response across patients administered either licensed trivalent inactivated influenza vaccine (TIV) or one of three doses (15, 45 or 135 μg) of trivalent recombinant baculovirus expressed hemagglutinin vaccines. | 3 Years

CONTACTS AND LOCATIONS:
Overall Officials: Amar Safdar, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- U.T.M.D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org